CLINICAL TRIAL: NCT04885088
Title: Smart Home Care of Cloud Base ECG on the Cardiotoxicity Prevention on the Cancer Patients.
Acronym: AI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ju-Chi Liu (Other)
Collaborators: Taipei Medical University WanFang Hospital (Other); Taipei Medical University Hospital (Other); Lotung Poh-Ai Hospital (Other)
Responsible Party: Sponsor-Investigator, Ju-Chi Liu, MD, PHD, Taipei Medical University Shuang Ho Hospital
Organization: Taipei Medical University Shuang Ho Hospital (Other)
Other Study IDs: ShuangHoH
Record Dates: First submitted 2021-05-09; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Artificial Intelligent; Cardiotoxicity; Cardiac Monitor; Cancer Treatment; ECG
Keywords: Artificial Intelligent; cardiotoxicity; Cardiac monitor; cancer treatment; ECG
MeSH Terms: conditions — Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Interventions: Device: Wisdom bracelet
  Other Names:
  control group (routine medical)
  Interventions: Device: Wisdom bracelet
- control: routine medical Non-invasive Wearable Device
  Interventions: Device: Wisdom bracelet

INTERVENTIONS:
Device: Wisdom bracelet — Wisdom bracelet

SUMMARY:
Thoracic malignancy is the most commonly diagnosed cancer worldwide.1,2 The incidence of thoracic malignancy has decreased in North America, but not in Asia, where it continues to show an increasing trend. A notable manifestation of the bimodal age distribution of thoracic malignancy has been observed in women. The occurrence of early-onset thoracic malignancy in the Asian population is earlier than that in the Western population, resulting in a higher incidence of thoracic malignancy in young Asian women. Moreover, the late onset age distribution of patients with thoracic malignancy in Asia (40-50 years) is earlier than that in Western countries (60-70 years), peaking at the age of 45-50 years in most women. The age-specific incidence rates of thoracic malignancy increase sharply until the menopausal stage.

Cardiovascular morbidity is higher among women with thoracic malignancy involving the thorax who had received radiotherapy (RT) compared with those not involving the thorax but receiving the same treatment. Thus far, the risks and time to onset of cardiac complications have been unclear in both young and old women. The proportion of young women with thoracic malignancy is higher in Asia than in Western countries. Furthermore, whether Asian women with thoracic malignancy are susceptible to RT remains unclear.

Anthracyclines are important therapeutic agents for breast cancer. Anthracycline-based regimens have similar or improved outcomes relative to the standard treatment regimen of cyclophosphamide, methotrexate, and fluorouracil. However, cardiotoxicity is a long-term toxicity associated with these regimens. The combined use of adjuvant anthracycline-based chemotherapy (CT) and RT may result in high cardiotoxicity. Nonetheless, no clear information on the effects of this combined therapy on the time to onset of both cardiac complications and cardiotoxicity is available. Furthermore, whether the cardiotoxicity of adjuvant RT and anthracycline-based CT is associated with age and ethnicity in women with thoracic malignancy remains unclear.

Therefore, cardiovascular disease is undoubtedly one of the most challenging health problems in the world. More efforts are needed to prevent and better control of this disease. Our proposed monitoring program is to use AI to monitor the basal value variation of personalized cardiovascular disease in cancer patients before and after chemoradiation. In the first year, our team focused on cardiotoxicity associated with cardiovascular disease models and cancer treatments. In the second year, we will apply knowledge in a clinical setting and calculate the severity of cardiac toxicity and its incidence and time response after cancer treatment. In the third year, high-risk groups will be identified to provide preventive intervention to reduce the risk of cancer-treatment related cardiotoxicity.

DETAILED DESCRIPTION:
This study is open, prospective study, multi-center, randomized controlled trial, unobtrusive research. This study is start on June 1 2021. And will include 400 patients who have just cardiotoxicity of adjuvant RT and anthracycline-based CT patients who diagnosis of Thoracic malignancy. And random allocation 200 experimental group (Non-invasive Wearable Device) and 200 control group (routine medical).

Ask whether the patients who meet the exclusion criteria are willing to participate in the screening (Screening), if they are willing to join and sign the consent of the subject, and after the patient's condition is stable, conduct an electrocardiogram (V0) before discharge from the hospital. On day 7 (±2 weeks), day 84 (±4 weeks), 168 days (±4 weeks), 252 days (±4 weeks), 336 days (±8 weeks) during routine clinical referral (V1-V5) Both are done once. The results of these two tests and other basic information of the patient, including Demography, Vital Signs, High, Weight, Medication, and European and Taiwan Cardiology Association recommended routine test results of high-risk patients, including Blood Chemistry Panel, NT-proBNP, Echocardiography, Myocardial Perfusion Scan, etc., will record the information of the logged-in subjects on the paper case report form. The CRF only displays the study number, and no subject is available. In addition to the examination of each return visit, the subjects also took the ECG bracelet home at the time of discharge (V0) and wore it every day. After the discharge, the ECG was measured every morning and evening, and their personal activity and sleep were collected. Relevant information. After the subject was discharged from the hospital, the subject tracked the date of all adverse events due to cardiovascular disease within one year, including: heart failure, restenosis due to blood vessel, and non-fatal myocardial infarction , To do blood vessel-related surgery again, and data on the occurrence of death.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 20-year-old
2. Patients who had received radiotherapy (RT) or anthracycline-based CT or cancer immunotherapy or Targeted Therapy
3. Diagnosis of Thoracic malignancy or breast cancer.
4. Willing to sign the consent form of the subject and cooperate with the return visit
5. Those who are admitted to the hospital and enter the general ward can receive the first ECG heart sound examination

Exclusion Criteria:

1. <20-year-old
2. Can't received radiotherapy (RT) or anthracycline-based CT or cancer immunotherapy or Targeted Therapy
3. Those who cannot perform the first examination after being admitted to the hospital and entering the general ward
4. It is impossible to measure the group of ECG and heart sounds. For example, when using Pacemaker, the ECG showed ventricular tachycardia (VT) and Dextrocardia on admission.
5. Patients who are bedridden and have difficulty in cooperating with return visits
6. Any subject that the physician believes is at high risk for future uncooperative tracking
7. Direct participants in this program

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age>=20,Physician diagnosed with Patients who had received radiotherapy (RT) or anthracycline-based CT or cancer immunotherapy or Targeted Therapy.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
death | Within a year
  death, divided into yes or no
heart failure | Within a year
  Come back to the hospital for heart failure (Judged by the physician) after discharge, divided into yes or no
Acute Coronary Syndrome, Coronary Artery Disease | Within a year
  Come back to the hospital for Acute Coronary Syndrome, Coronary Artery Disease (Judged by the physician) after discharge, divided into yes or no
Myocarditis | Within a year
  Come back to the hospital for Myocarditis (Judged by the physician) after discharge, divided into yes or no

SECONDARY OUTCOMES:
Arrhythmia | Within a year
  Re-hospitalization for Arrhythmia (Judged by the physician) after discharge, divided into yes or no
Valvular Heart Disease | Within a year
  Re-hospitalization for Valvular Heart Disease (Judged by the physician) after discharge, divided into yes or no
Physician adjusts medicine | Within a year
  According to the medicine order issued by the doctor, if there is any adjustment of the medicine, make a record,divided into yes or no
Physician arranges examination early | Within a year
  If the doctor has arranged to do Cardiac ultrasound or stress & redistribution myocardial perfusion scan with SPECT During non-table period, divided into yes or no
Compliance | Within a year
  Judged by the physician, when the patient returns to the consultation, the patient is asked about the compliance with the drug in the past, divided into yes or no
Medical cost | Within a year
  The sum of all medical and health insurance expenses of the patient in the past year

CONTACTS AND LOCATIONS:
Overall Officials: Ju-Chi Liu, PHD, MD, Study Chair — Taipei Medical University Shuang Ho Hospital

IPD SHARING:
Plan to Share IPD: No